CLINICAL TRIAL: NCT05249738
Title: Detection of Tongue Edema Caused by Intubation Tube in Intensive Care Unit Patients by Ultrasonography
Brief Title: Tongue Edema Caused by Intubation Tube in Intensive Care Unit Patients
Status: Completed | Type: Observational
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Ozkan Onal, Associate Professor, Selcuk University
Other Study IDs: 02.10.2019-241
Record Dates: First submitted 2022-02-11; First posted 2022-02-22 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Tongue Edema; Tongue Enlarged; Mechanical Ventilation Complication; Intubation Complication
Keywords: ultrasonography; endotracheal intubation tube; complication; drugs; tongue edema
MeSH Terms: conditions — Macroglossia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Group: Patients followed up with a mechanical ventilator for 4 days or longer were included in the study group.
  Interventions: Diagnostic Test: Measuring tongue cross-sectional area by submental ultrasonography
- Control Group: Patients followed up with mechanical ventilation for 3 days or less were included in the control group.
  Interventions: Diagnostic Test: Measuring tongue cross-sectional area by submental ultrasonography

INTERVENTIONS:
Diagnostic Test: Measuring tongue cross-sectional area by submental ultrasonography — The tongue cross-sectional areas of both groups were measured with submental ultrasonography to detect tongue edema.

SUMMARY:
Tongue edema (TE) is an enlargement of the tongue that can be noticed with the naked eye and protrudes from the mouth. Endotracheal intubation tube, which can exert high pressure on the tongue for a long time, may cause TE. This study was aimed to detect TE, which may develop due to long-term pressure application of the intubation tube to the tongue, in patients hospitalized in the intensive care unit (ICU) who underwent endotracheal intubation by submental ultrasonography (USG) method.

DETAILED DESCRIPTION:
Tongue edema (TE) is an enlargement of the tongue that can be noticed with the naked eye and protrudes from the mouth. Endotracheal intubation tube, which can exert high pressure on the tongue for a long time, may cause TE. This study was aimed to detect TE, which may develop due to long-term pressure application of the intubation tube to the tongue, in patients hospitalized in the intensive care unit (ICU) who underwent endotracheal intubation by submental ultrasonography (USG) method.

ELIGIBILITY:
Inclusion Criteria:

Patients aged between 18-65 years Patients who underwent endotracheal intubation and were admitted to the intensive care unit on the 0th day of intubation and patients who underwent endotracheal intubation during follow-up in the intensive care unit and were followed up on a mechanical ventilator -

Exclusion Criteria:

Patients under the age of 18 and over the age of 65 Patients who had a history of maxillofacial trauma, tongue surgery, head and neck malignancy, radiotherapy to the head and neck region, congenital anomalies of the tongue base and floor of the mouth Patients who were admitted to the intensive care unit due to allergy-anaphylaxis

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients who underwent endotracheal intubation in the Anesthesiology and Reanimation intensive care unit were followed up on a mechanical ventilator were included in the study after obtaining informed consent from their legal representatives.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Detection of tongue edema by ultrasonography | The patients' tongue cross-sectional areas were measured by submental ultrasonograph on the 0th day of endotracheal intubation and 4th day of follow-up on a mechanical ventilator. The difference between the two measurements was evaluated as tongue edema.
  Primary outcome was tongue edema which is likely to develop due to the pressure exerted by endotracheal intubation tube on the tongue, by submental ultrasonography in patients who were followed up on mechanical ventilation for a long time.

SECONDARY OUTCOMES:
The effect of drugs applied in the intensive care unit on the development of tongue edema | The patients' tongue cross-sectional areas were measured by submental ultrasonograph on the 0th day of endotracheal intubation and 4th day of follow-up on a mechanical ventilator. The difference between the two measurements was evaluated as tongue edema.
  Secondary outcome was tongue edema which is likely to develop due to the drugs applied in the intensive care unit by submental ultrasonography.

OTHER OUTCOMES:
The effect of the inner diameter of endotracheal intubation tube on the development of tongue edema. | The patients' tongue cross-sectional areas were measured by submental ultrasonograph on the 0th day of endotracheal intubation and 4th day of follow-up on a mechanical ventilator. The difference between the two measurements was evaluated as tongue edema.
  The exploratory outcome was tongue edema which is likely to develop due to the intubation tube with a large inner diameter.

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University, Konya, Selcuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Study protocol, statistical analysis plan and raw data can be shared individual if there is a valid reason.

REFERENCES:
- [Result] Onal M, Colpan B, Elsurer C, Bozkurt MK, Ozturk M, Onal O, Turan A. Can Tonsillar Retractor-Induced Tongue Edema Be a New Complication in Pediatric Patients Undergoing Tonsillectomy Detected by Ultrasonography? A Prospective, Case-Controlled, Observational Study. Ear Nose Throat J. 2022 Jan;101(1):42-47. doi: 10.1177/0145561320934918. Epub 2020 Jul 7. PMID 32633658
- [Result] Onal M, Colpan B, Elsurer C, Bozkurt MK, Onal O, Turan A. Is it possible that direct rigid laryngoscope-related ischemia-reperfusion injury occurs in the tongue during suspension laryngoscopy as detected by ultrasonography: a prospective controlled study. Acta Otolaryngol. 2020 Jul;140(7):583-588. doi: 10.1080/00016489.2020.1743353. Epub 2020 Mar 30. PMID 32223688
- [Derived] Bayram HH, Onal O, Akpinar S, Onal M, Aslanlar E, Ozturk M. Detection of tongue edema caused by endotracheal intubation tube in ICU patients by ultrasonography: a prospective, observational, clinical study. J Clin Monit Comput. 2024 Jun;38(3):721-729. doi: 10.1007/s10877-023-01123-0. Epub 2024 Jan 19. PMID 38240918